CLINICAL TRIAL: NCT04455321
Title: The Effect of Suture Materials With Different Absorption Times on Isthmocele: Prospective Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Selçuk Yetkinel, MD., Baskent University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KA19/170
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Suture, Complication; Istmocel
Keywords: rapid; suture material; istmocel
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: Rapid vicryl will used in study group and vicryl will used in control group for uterine closure in cesarean section.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicryl (Active Comparator): Single layer locked uterine closure with vicryl suture material
  Interventions: Procedure: Suture materials effect on istmocel
- rapide vicryl (Experimental): Single layer locked uterine closure with rapide vicryl suture material
  Interventions: Procedure: Suture materials effect on istmocel

INTERVENTIONS:
Procedure: Suture materials effect on istmocel — Effect of suture materials with different absorption times on istmocel

SUMMARY:
This study aims to investigate the effect of suture materials with different absorption times on istmocel.

ELIGIBILITY:
Inclusion Criteria:

* primary cesarean section
* single pregnancy
* 18-45 age

Exclusion Criteria:

* Diabetes mellitus disease
* inflammatory bowel disease
* systemic lupus erythematosus disease
* rheumatoid arthritis disease
* previous uterine surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Istmocel | Six months
  Istmocel area measurement with saline-infusion ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Adana Dr. Turgut Noyan Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No